CLINICAL TRIAL: NCT04986839
Title: PAIR (Paracetamol and Ibuprofen Research) Study: A Randomised Controlled Trial Comparing IV Paracetamol With IV Ibuprofen in the Management of Haemodynamically Significant Patent Ductus Arteriosus
Brief Title: PAIR (Paracetamol and Ibuprofen Research) Pilot Trial
Acronym: PAIR
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B01039
Record Dates: First submitted 2021-07-19; First posted 2021-08-03 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: The study involves two-arm parallel assignment where one group receives standard treatment (Ibuprofen) and the other group receives investigational medicinal product (Paracetamol) to treat Patent Ductus Arteriosus
Who Masked: Outcomes Assessor
Masking Description: Infants will be randomized. Outcome assessor of the treatment will be blinded to the trial participants. No allocation concealment is done.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen (Active Comparator): Standard treatment arm which will provide the comparator arm to the proposed new treatment. This is routine standard of practice
  Interventions: Drug: Ibuprofen injection
- Paracetamol (Experimental): To study the efficacy of Paracetamol (proposed new treatment) in treating hsPDA in comparison to Ibuprofen (current standard treatment) in preterm infants
  Interventions: Drug: Paracetamol injection

INTERVENTIONS:
Drug: Paracetamol injection — Intravenous Paracetamol
  Other Names: Acetaminophen
  Arms: Paracetamol
Drug: Ibuprofen injection — Intravenous Ibuprofen
  Other Names: Brufen
  Arms: Ibuprofen

SUMMARY:
Presence of Patent Ductus Arteriosus is detrimental to an infant born prematurely. The primary objective is to study the efficacy of Paracetamol (proposed new treatment) in treating haemodynamic significant Patent Ductus Arteriosus (hsPDA) in comparison to Ibuprofen (current standard treatment) in preterm infants. Outcome of such treatment will check on the conversion of hsPDA to non-hsPDA. All preterm infants (born at <32 weeks gestational age or birth weight < 1500 grams) with haemodynamically significant patent ductus arteriosus (hsPDA) who are ≤ 28 days old will be included over 2 years. Sample size 32. Secondary outcomes of this study will compare

1) BPD (broncho-pulmonary dysplasia) free survival at 36 weeks post menstrual age (PMA), 2) incidence of complications of prematurity in each group and 3) to record any evidence of adverse effects with Paracetamol or Ibuprofen.

DETAILED DESCRIPTION:
Patent Ductus Arteriosus (PDA) is present in 40-60 percent of preterm infants. A persistent PDA with a large left to right ductal shunt may be 'haemodynamically significant' (hsPDA) resulting in pulmonary hyper-perfusion and systemic hypo-perfusion. The association of a PDA with an increased incidence of pulmonary haemorrhage, bronchopulmonary dysplasia and prolonged need for ventilatory support is ascribed to pulmonary hyper-perfusion, whereas necrotising enterocolitis, renal failure, cerebral haemorrhage, and periventricular leukomalacia are consequences of systemic hypo-perfusion. In the United Kingdom, Ibuprofen (a non-steroidal anti-inflammatory drug, NSAID) is used to treat hsPDA in preterm babies. Paracetamol has come up recently as a promising alternative with fewer side effects and has been used in the management of PDA with promising results. However, the current available body of evidence is considered to be of moderate to low quality and hence its effectiveness and safety profile is not fully established in this patient population. The primary objective is to study the efficacy of IV paracetamol in treating hsPDA in comparison to IV ibuprofen in preterm infants born at less than 32 weeks' gestation OR less than 1500 grams birth weight.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age - <32 weeks OR birth weight < 1500 grams
* Postnatal age ≤ 28 days
* Meets criteria for hsPDA
* Clinician's decision to treat PDA

Exclusion Criteria:

* Contraindication for administration of Ibuprofen (cyclooxygenase-inhibitors) or Paracetamol, such as: active bleeding (e.g. intracranial or gastrointestinal haemorrhage), thrombocytopenia (<50x109/L), renal failure (raised creatinine (>100 micromole/l) or oliguria (<0.5 mL/kg/hour), known or suspected necrotising enterocolitis, any gastric or intestinal perforation, pre-treatment abnormal liver function tests (ALT > upper normal limit of the reference range, Bilirubin > National Institute of Clinical Excellence exchange phototherapy level).
* Previous use of Ibuprofen or Paracetamol prior to randomisation.
* Persistent pulmonary hypertension (ductal right-to-left shunt ≧33% of cardiac cycle).
* Congenital heart defect, other than PDA or Patent Foramen Ovale (PFO).
* Life-threatening congenital birth defects.
* Chromosomal abnormalities and/or congenital anomalies associated with abnormal neurodevelopment.

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Conversion of haemodynamically significant PDA (hsPDA) to non-hsPDA | 3 days
  Efficacy of Paracetamol (proposed new treatment) in treating hsPDA in comparison to Ibuprofen (current standard treatment) in preterm infants. The diagnosis of hsPDA will be made in the presence of supportive clinical signs and at least three of the following echocardiogram indices:
  i) PDA diameter ≥2.0 mm in 2D ii) Ductal flow pattern ('growing' pattern or pulsatile with Vmax/Vmin ≥ 2) iii) Retrograde post ductal aortic/coeliac/SMA (superior mesenteric artery) diastolic flow iv) LA/Ao ratio (left atrium:Aorta) ≥ 2 v) LVO (Left ventricular output) ≥ 300 ml/kg/min vi) Mitral valve E/A ratio ≥ 1
  An echocardiogram will be carried out within 72 hours of the last dose and PDA will be classified as non-hsPDA based on the following criteria - PDA closed OR any two of the following three parameters i) Reduction of PDA diameter >50% (2D) ii) Restrictive or closing Ductal flow pattern iii) LA: Ao ratio < 1.5

SECONDARY OUTCOMES:
Broncho-pulmonary dysplasia (BPD) free survival at 36 weeks post menstrual age (PMA) | Age up to 36 weeks PMA
  BPD free survival at 36 weeks PMA
Incidence of complications of prematurity in each group | Age up to 36 weeks PMA
  1. Necrotising enterocolitis (NEC, Bell stage ≥IIa)
  2. Significant intraventricular haemorrhage ( IVH) grade 3/4)
  3. Retinopathy of Prematurity (ROP) requiring treatment
To record any evidence of adverse effects with Paracetamol or Ibuprofen | Within 7 days of starting the trial medications
  . a) Renal impairment (elevated urea and creatinine > upper limit of normal range) b) Hepatic impairment (elevated liver enzymes ALT or Aspartate transaminase (AST) > upper limit of normal) c) Significant gastrointestinal or non-gastrointestinal bleeding requiring intervention

CONTACTS AND LOCATIONS:
Overall Officials: Arin Mukherjee, MRCPCH, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mukherjee A, Gupta A, Fullwood C, Gottstein R. Paracetamol or ibuprofen? A pilot study comparing rescue therapy for PDA in preterm infants within the first month. Front Pediatr. 2026 Jan 2;13:1717284. doi: 10.3389/fped.2025.1717284. eCollection 2025. PMID 41550606

DOCUMENTS (2):
  • Study Protocol (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT04986839/Prot_000.pdf
  • Informed Consent Form (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT04986839/ICF_001.pdf